## Lavage of the Uterine Cavity for Diagnosis of Ovarian Cancer

NCT03606486

Date: 12/4/23

## Lavage of the Uterine Cavity for Diagnosis of Ovarian Carcinomas Statistical Analysis Plan

Comparison of mutation frequencies, mutation burden, and variant allele fraction (VAF) across groups of individuals was performed by Mann-Whitney U test. Correlations were tested with Spearman's rank test. Associations between categorical variables were tested with Fisher exact test. Two logistic regression models were constructed, one including the standard ovarian cancer risk variables (age and CA-125) and an exploratory model including age, CA-125 and TP53 mutation burden. The models equated the relationship between variables with the occurrence of ovarian cancer to estimate beta coefficients with 95% confidence intervals. Due to a heavy right-tailed distribution, CA-125 was log transformed. Age and TP53 mutation burden were presented as a per standard deviation (SD) increase. All tests were two-sided at an alpha level (type 1 error rate) of 0.05. Statistical analyses were performed with SPSS version 26, R version 4.1.1, and Stata 16.